CLINICAL TRIAL: NCT02776670
Title: Clinical Evaluation Following Use of SYSTANE® BALANCE in Subjects With Lipid-Deficient Dry Eye
Brief Title: Clinical Outcomes Following Treatment With SYSTANE® BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXB107-P001
Record Dates: First submitted 2016-05-17; First posted 2016-05-18 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Propylene Glycol; Ophthalmic Solutions; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYSTANE BALANCE (Experimental): Propylene glycol, 0.6% eye drops, 1 drop in each eye 4 times per day for 35 days
  Interventions: Other: Propylene glycol, 0.6% eye drops
- REFRESH OPTIVE (Active Comparator): Lubricant eye drops, 1 drop in each eye 4 times per day for 35 days
  Interventions: Other: Lubricant eye drops

INTERVENTIONS:
Other: Propylene glycol, 0.6% eye drops
  Other Names: SYSTANE® BALANCE
  Arms: SYSTANE BALANCE
Other: Lubricant eye drops
  Other Names: REFRESH OPTIVE® Advanced
  Arms: REFRESH OPTIVE

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of SYSTANE® BALANCE compared to REFRESH OPTIVE® Advanced in subjects with lipid-deficient dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to attend all study visits;
* Must sign an informed consent form;
* Best-corrected visual acuity (BCVA) of 55 letters or better in each eye as assessed using an early treatment diabetic retinopathy study (ETDRS) chart;
* Willing to take study products as directed for entire study;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, plan to become pregnant during the study, breast feeding, or not using adequate birth control methods;
* Contact lens use within 30 days prior to Screening Visit, or unwilling to avoid contact lens use during the course of the study;
* Use of medication excluded by the protocol;
* Diseases, illnesses, infections, or ocular abnormalities excluded by the protocol;
* Ocular surgeries or procedures excluded by the protocol;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Manager, PLS, Study Director — Alcon, a Novartis Company

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 14 study centers located in Australia (2), Taiwan (1), Singapore (1), United Kingdom (1) and the US (9).
Pre-assignment Details: Of the 308 enrolled, 77 were exited as screen failures prior to randomization. This reporting group includes all randomized and treated subjects (231).
Period: Overall Study
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE
Started (Randomized and treated) | 117 | 114
Full Analysis Set (FAS) (All randomized subjects who had at least 1 post-baseline primary endpoint (ie, TFBUT) assessment.) | 117 | 114
Per Protocol Analysis Set (PPS) (Subjects in FAS who satisfied all inclusion/exclusion criteria and had no major protocol deviations) | 115 | 113
Safety Analysis Set (All subjects exposed to post-randomization study treatment) | 117 | 114
Completed (All subjects who completed the study whether on study treatment or not) | 117 | 108
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other - Reason not given | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were randomized to one of the study treatment arms (Randomized Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE | Total
Number analyzed (Participants) | 117 | 114 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (14.70) | 55.6 (16.35) | 56.2 (15.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 92 | 182
  Male | 27 | 22 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 25 | 27 | 52
  Black or African American | 6 | 7 | 13
  Multiracial | 1 | 1 | 2
  White | 81 | 76 | 157
  Other | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Tear Film Break-Up Time (TFBUT) at Day 35
Description: TFBUT (the time required for dry spots to appear on the surface of the eye after blinking) was assessed with a fluorescein strip and measured in seconds. Using a stopwatch, the investigator measured the time from the last blink until one or more black (dry) spots appeared in the precorneal tear film. The longer it takes, the more stable the tear film. A positive number change from baseline indicates improvement. Only one eye (analysis eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 35
Population: Per Protocol Analysis Set. At each time point, only subjects with a value at both Baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE
Number analyzed (Participants) | 115 | 110
seconds | 0.999 (1.9439) | 0.864 (1.6198)
Statistical Analysis 1: Comparison: SYSTANE BALANCE vs REFRESH OPTIVE; Test type: Non-Inferiority — Noninferiority was deemed established if the lower limit of the 95% CI (equivalent to the 1-sided 97.5% CI) for the adjusted estimate of the difference (Systane Balance-Refresh Optive Advanced/Optive Plus) was above the noninferiority margin of -1.0 second; p < 0.0001, Mixed model repeated measures (MMRM) — p-value for testing noninferiority of Systane Balance with respect to Refresh Optive Advanced/Refresh Optive Plus is calculated for predefined noninferiority margin of -1.0 second; Mean Difference (Final Values) = 0.130, 95% CI 2-sided [-0.341 to 0.601]

2. Secondary Outcome: Change From Baseline in TFBUT at Day 35
Description: as for outcome 1
Time Frame: Baseline (Day 0), Day 35
Population: Full Analysis Set. At each time point, only subjects with a value at both Baseline and that time point are included.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE
Number analyzed (Participants) | 117 | 110
seconds | 0.985 (0.1651) | 0.867 (0.1702)
Statistical Analysis 1: Comparison: SYSTANE BALANCE vs REFRESH OPTIVE; Test type: Superiority; p = 0.310, MMRM; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [-0.349 to 0.585]

3. Secondary Outcome: Lipid Layer Thickness (LLT) Area Under the Curve (AUC120) at Day 35
Description: LLT was measured using the LipiView® Ocular Surface Interferometer, an ophthalmic imaging device intended for use in adult patients to capture, archive, manipulate and store digital images of specular (interferometric) observations of the tear film, which can be visually monitored and photographically documented. Using these images, the LipiView® Interferometer measures the absolute thickness of the tear film lipid layer.
Time Frame: Day 35
Population: Area under the curve (AUC) lipid layer thickness (LLT) was removed from formal analysis as a secondary endpoint via amendment of the standalone Statistical Analysis Plan (SAP) due to a large proportion of data that were above the limit of detection.
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change From Baseline in Global Ocular Discomfort Visual Analog Scale (VAS) Score at Day 35
Description: Ocular discomfort frequency and severity (each graded on a separate 100-units scale) were assessed using a visual analog scale (VAS). Frequency score was in response to the question 'how often your eyes felt uncomfortable during the past week' ranging from 'Rarely' to 'All the time.' Severity score was in response to the question 'how uncomfortable your eyes felt during the past week' ranging from 'Very mildly uncomfortable' to 'Very severely uncomfortable.' The Global Ocular Discomfort Score, ranging from 0 to 100, was calculated for the given visit, as the square root of the product of the ocular discomfort frequency score multiplied by the ocular discomfort severity score. Improvement results in a reduction of the ocular discomfort frequency or severity, or both, translating into a reduction of the resulting Global Ocular Discomfort score as compared to baseline. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0), Day 35
Population: Full Analysis Set. At each time point, only subjects with a value at both Baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE
Number analyzed (Participants) | 117 | 110
units on a scale | -9.9 (25.26) | -8.8 (26.11)
Statistical Analysis 1: Comparison: SYSTANE BALANCE vs REFRESH OPTIVE; Test type: Superiority; p = 0.618, MMRM; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-6.4 to 4.7]

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) through study completion, an average of 35 days. Adverse Events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Description: This analysis population includes all subjects exposed to post-randomization study treatment (Safety Analysis Set), as treated. Two subjects were randomized to one of the study drugs but received the other instead. Specifically, one subject was randomized to REFRESH OPTIVE®, but received SYSTANE® BALANCE instead; and a different subject was randomized to SYSTANE® BALANCE, but received REFRESH OPTIVE® instead.
Groups:
- SYSTANE BALANCE: All subjects exposed to SYSTANE® BALANCE
- REFRESH OPTIVE: All subjects exposed to REFRESH OPTIVE®
Arm/Group | SYSTANE BALANCE | REFRESH OPTIVE
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/117 | 1/114
Other Adverse Events (participants affected / at risk) | 6/117 | 13/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYSTANE BALANCE (N=117) | REFRESH OPTIVE (N=114)
Abscess neck (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SYSTANE BALANCE (N=117) | REFRESH OPTIVE (N=114)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 4
Conjunctival hyperaemia (Eye disorders) | 1 | 3
Eye irritation (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 0 | 3
Posterior capsule opacification (Eye disorders) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 3
Vital dye staining cornea present (Investigations) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT02776670/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02776670/SAP_001.pdf